CLINICAL TRIAL: NCT01964196
Title: ASP1517 Phase 2 Clinical Trial -A Multi-center, Randomized, Parallel Groups, Placebo-controlled, Double-Blind Study of ASP1517 for the Treatment of Anemia in Chronic Kidney Disease Patients Not on Dialysis-
Brief Title: ASP1517 Phase 2 Clinical Trial - Double-Blind Study of ASP1517 for the Treatment of Anemia in Chronic Kidney Disease Patients Not on Dialysis-
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1517-CL-0303
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Anemia in Chronic Kidney Disease Patients Not on Dialysis
Keywords: Chronic Renal Failure; Renal anemia; ASP1517
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASP1517 low dose group (Experimental): Oral
  Interventions: Drug: ASP1517
- ASP1517 middle dose group (Experimental): Oral
  Interventions: Drug: ASP1517
- ASP1517 high dose group (Experimental): Oral
  Interventions: Drug: ASP1517
- Placebo group (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP1517 — Oral administration
  Arms: ASP1517 high dose group; ASP1517 low dose group; ASP1517 middle dose group
Drug: Placebo — Oral
  Arms: Placebo group

SUMMARY:
This study is to evaluate the safety and the dose-response of ASP1517 in the treatment of anemia in non-dialysis Chronic Kidney Disease (CKD) patients when ASP1517 is applied intermittently.

DETAILED DESCRIPTION:
To evaluate the safety and the dose-response of ASP1517 on Hemoglobin (Hb) correction in the treatment of anemia in non-dialysis Chronic Kidney Disease (CKD) patients when ASP1517 is applied intermittently. Patients will receive ASP1517 three times a week (TIW) for first 6weeks. Patients may have the second-randomization to TIW dosing or once-a-week (QW) dosing at Week 6, 8, 10, 12, 14 or 16 if patients meet the criteria.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease with an estimated glomerular filtration rate (as calculated by the Japanese GFR estimation equation) of =<89 mL/min/1.73 m2, and not required dialysis for 3 months since study completion
* The mean of two Hb values at screening test and Hb test (at least one week apart form the screening test) is <10.0 g/dL, with a difference of ≤1.0 g/dL between the two values
* Both TSAT>=5% and ferritin >=30 ng/mL at screening test
* Serum folate ≥4.0 ng/mL and Vitamin B12 ≥180 pg/mL at screening test

Exclusion Criteria:

* Proliferative retinopathy, age-related macular degeneration, retinal vein occlusion and/or macular edema that is considered to require treatment
* Immunological disease with severe inflammation as assessed by the Investigator; even if the inflammation is in remission, the subject is excluded (e.g. lupus erythematosus, rheumatoid arthritis, Sjogren's syndrome, celiac disease, etc).
* Having a history of gastric/intestinal resection considered influential on the absorption of the drug in the gastrointestinal tract or evidence of active gastroparesis.
* Uncontrollable hypertension (more than one third blood pressure values of diastolic BP >100 mmHg within 16 weeks prior to screening test including)
* Congestive heart failure (NYHA classification III or higher)
* Having a history of hospitalization for stroke, myocardial infarction or lung infarction within 24 weeks before screening test
* Positive for any of the following: anti-hepatitis C virus antibody (anti-HCV Ab); hepatitis B surface antigen (HBsAg); or human immunodeficiency virus (HIV)
* Anemia other than anemia due to low/absent renal production of EPO (e.g., iron deficiency anemia, hemolytic anemia, pancytopenia, etc)
* Using ESA, anabolic androgenic steroid, testosterone enanthate or mepitiostane within 6 weeks before screening test

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2015-07-06 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of rise in Hb (g/dL/week) at Week 6 | Baseline and at 6 weeks after dosing

SECONDARY OUTCOMES:
Percentage of cumulative number of responder patients | for 28 weeks after dosing
  responder is defined as a Hb ≥10.0 g/dL and an increase in Hb by ≥1.0 g/dL
Percentage of visits at which patients maintain Hb between 10.0-12.0 g/dL after achieving Hb ≥10.0 g/dL for each patients | for 28 weeks after dosing
Percentage of patients who maintain Hb between 10.0-12.0 g/dL at each visit | Before and Week-2, -3, -4, -6, -8, -10, -12, -14, -16, -18, -20, -22, -24 and -28
Change from baseline in Hb | Before and Week-2, -3, -4, -6, -8, -10, -12, -14, -16, -18, -20, -22, -24 and -28
Safety assessed as the incidence of adverse events, vital signs, 12-lead ECGs and lab-tests | for 28 weeks after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Akizawa T, Iwasaki M, Otsuka T, Reusch M, Misumi T. Roxadustat Treatment of Chronic Kidney Disease-Associated Anemia in Japanese Patients Not on Dialysis: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial. Adv Ther. 2019 Jun;36(6):1438-1454. doi: 10.1007/s12325-019-00943-4. Epub 2019 Apr 5. PMID 30953333
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=397